CLINICAL TRIAL: NCT06959992
Title: Evaluating the Efficacy of Virtual Support Groups Fostering Resilience for Gender Diverse People: a Randomized Clinical Trial in the Metaverse
Brief Title: Developing Resilience in Transgender and Nonbinary Individuals - Exploring the Impact of Social Challenges in the Metaverse
Acronym: RESILIDENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Responsible Party: Principal Investigator, Cezar Giosan, Associate Professor of Psychology, University of Bucharest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123/01.10.2024
Record Dates: First submitted 2025-04-17; First posted 2025-05-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Resilience,Psychological; Well-Being, Psychological; Self-Compassion
Keywords: Metaverse; Gender minorities; Support groups; Resilience; Well-being; Randomized clinical trial; Self-compassion
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metaverse group (Experimental): Immersive online environment
  Interventions: Behavioral: Metaverse group
- Standard asynchronous online group (Active Comparator): Online environment
  Interventions: Behavioral: Online asynchronously
- Waitlist (No Intervention): Control

INTERVENTIONS:
Behavioral: Metaverse group — The activities will be conducted in a Metaverse platform with immersive features. Each session is divided into two parts (~2 hours duration). First, a specific social context will be represented (environmental features and static avatars) and a microaggression scenario (adapted for the chosen context) will be described. Participants are engaged in the conversation by the moderator in order to identify various psychological manifestations regarding the context (according to the SORC model) and to come up with solutions for the main, model avatar (part of the research team). Second, the debriefing part of the session will allow participants to talk about their own experiences alongside specific self-compassionate exercises. Repeated measurements will be required: pre-intervention, mid-intervention, post-intervention and at follow-up (after 3 months).
  Arms: Metaverse group
Behavioral: Online asynchronously — The activities will be conducted asynchronously in an online platform where participants will be guided by the moderator through the same type of activities. First, a social context with specific microaggressions will be presented in a text format followed by the same requirements for participants (identifying various psychological manifestations regarding the context and coming up with solutions for the problematic situation). Second, participants will have the transcripts of several self-compassionate exercises to be done independently. A discussion forum will also require their active engagement. Repeated measurements will be required pre-interventions, mid-intervention, post-intervention and at follow-up (3 months).
  Arms: Standard asynchronous online group

SUMMARY:
The goal of this clinical trial is to test the effectiveness of conducting a support group in the Metaverse designed to develop and/or improve resilience in gender diverse people. By exploring the impact of different social challenges in a virtual environment, the main question it aims to answer is whether this approach on conducting support group sessions with gender diverse people will strengthen their resilience and associated abilities (self-compassion) compared to a control group and a waitlist.

DETAILED DESCRIPTION:
The gender diverse population is inclined toward online expression as a way to connect with the community and to explore ways of handling stigma from harsh environments that they live in. The potential beneficial effects of conducting a support group to build resilience and self-compassion, with members from the gender minority community in a virtual environment, allowing the expression of gender identity through avatar customization and social interaction are being tested in the form of a Randomized Clinical Trial (RCT). There are three conditions: the virtual group (enrolling in a Metaverse platform with immersive features), the standard group (enrolling in an online forum platform) and the waitlist group.

The study is a between-subjects design with three arms and involves comparisons between pre-intervention, post-intervention and follow-up between: (a) Initial psychological states of the participants, (b) Mid-session, (c) After the support group sessions and (d) At follow-up (3 months). Participants will be randomly allocated to one of the three experimental arms.

For small-medium effect sizes assumed (f = 0.20), 3 groups and 4 measurements in time (pre- and post-intervention and one follow-up), a repeated measure analyzing between-within factors a minimum of 45 participants (total sample size) are needed. A target of 123 people (41 per group) has been set to allow for potential dropouts (~20%).

The group sessions should be re-run several times as the chosen Metaverse platform and the general recommendations for conducting support groups limit the number of participants to 7-8 people/group.

ELIGIBILITY:
Inclusion Criteria:

* Gender diverse people with a stable gender-identity or questioning

Exclusion Criteria:

* Formally diagnosed with a mental disorder
* Not being part of the gender minority population
* Younger than 18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Gender-affirmation | Up to 5 months
  Assessing changes in levels of comfort and satisfaction related to gender identity with The Psychological Gender Affirmation Scale which contains 5 items, ranging from 1 - Not at all to 5 - Extremely. Higher scores indicate better outcomes.
Resilience | Up to 5 months
  Assessing changes in resilient attitudes from a general perspective with the Brief Resilience Scale (6 items on a 5-point Likert response scale, ranging from 1 - Strongly disagree to 5 - Strongly agree) and from a specific view of gender minority resilience with the Gender Minority Stress and Resilience Measure. Only the resilience items will be selected from the 58-items scale (5 items for Community connectedness and 8 items for Pride). Responses range from 0 - Strongly disagree to 4 - Strongly agree. Higher scores indicate better outcomes.
Stress and mental health correlates | Up to 5 months
  Assessing changes in perceived distal (Discrimination, Rejection and Victimization - 17 items) and proximal stress factors (Non-affirmation of gender identity, Internalized transphobia, Nondisclosure and Negative future expectations - 28 items) with the Gender Minority Stress and Resilience Measure (selecting only stress-related items) and in mental health symptoms with the Depression, Anxiety, Stress Scale (DASS), containing 21 items. Higher scores mean worse outcomes.
Coping mechanisms | Up to 5 months
  Assessing changes in approached coping mechanisms with the Trans and Nonbinary Coping Measure containing 28 items and 6 subscales with both adaptive and maladaptive types of coping, on a 5-point Likert scale (1 - I do not do this to 5 - I almost always do this). Scoring significance depends on the nature of the coping mechanisms.
Self-compassion | Up to 5 months
  Assessing changes in self-compassionate attitudes with the Short Form of the Self-Compassion Scale, containing 12 items on a 5-point Likert response scale ranging from 1 - Almost never to 5 - Almost always. Higher scores mean better outcomes.
Social support | Up to 5 months
  Assessing changes in perceived social support with the Multidimensional Scale of Perceived Social Support, containing 12 items on a 7-point Likert response scale (ranging rom 1 - Very strongly disagree to 7 - Very strongly agree). Higher scores mean better outcomes.
Positive gender identity characteristics | Through study completion, an average of 3 months
  Assessing changes in positive characteristics of gender identity with the Transgender Positive Identity Measure with 24 items with a 7-point Likert response scale (ranging from 1 - Strongly disagree to 7 - Strongly agree).

SECONDARY OUTCOMES:
Mood changes | Through study completion, an average of 3 months
  Short mood check questions for the beggining and end of the sessions with items from The World Health Organization-Five Well-Being Index (6-point Likert scale).
Attitudes toward self | Up to 5 months
  Changes in self-focused attention specific to gender minorities with the Gender Identity Reflection and Rumination Scale, containing 15 items on a 4-point Likert scale (1 - almost never to 4 - almost always). Higher scores for reflection mean better outcomes.
Assertive attitude | Up to 5 months
  Changes in assertiveness are assessed with the Short Form of the Simple Rathus Assertiveness Scale, with 19 items on a 6-point Likert response format (1 - very unlike me to 6 - very much like me). Higher scores mean better outcomes.
Self-efficacy | Up to 5 months
  Assessing enhacement in self-efficay with the General Self-Efficacy Scale with 10 items on a 4-point Likert scale (1 - Not true at all to 4 - Exactly true). Higher scores mean better outcomes.

OTHER OUTCOMES:
Gender dysphoria | Baseline
  Gender dysphoric symptoms are assessed pre-intervention (at baseline) to establish an initial level of gender-dysphoria for participants with the Gender Preoccupation and Stability Questionnaire containing 14 items with a 5-point response Likert scale. Higher scores mean increased gender dysphoria.
Psychiatric problems | Baseline
  The DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure is used for a primary screening process at baseline to identify potential elevated psychiatric problems. Higher scores mean worse mental health conditions.
Microaggressions | Baseline
  Past experiences of microaggressions are assessed with two scales, one for binary transgender participants (Gender Identity Microaggressions Scale) containing 14 items, and one for nonbinary transgender participants (The Nonbinary Gender Microaggressions) Scale containing 23 items. Higher scores mean negative experiences with microaggresions.

CONTACTS AND LOCATIONS:
Overall Officials: Cezar Giosan, PhD, Principal Investigator — University of Bucharest
Locations (1):
- University of Bucharest, Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No